CLINICAL TRIAL: NCT00059878
Title: A Prospective, Randomized, Double-Blind, Multicenter Pilot Study Of The Safety And Efficacy Of Interferon Gamma- 1b (IFN-y 1b) Plus Voriconazole Versus Placebo Plus Voriconazole In The Treatment Of Invasive Aspergillosis And Other Filamentous Fungal Infections
Brief Title: Voriconazole With or Without Interferon Gamma in Treating Patients With Aspergillosis or Other Fungal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000298887; NCI-03-C-0111
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-07

CONDITIONS: Infection; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: infection; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Infections | interventions — Interferon-gamma; Voriconazole

INTERVENTIONS:
Biological: recombinant interferon gamma
Drug: voriconazole

SUMMARY:
RATIONALE: Antifungals such as voriconazole may be effective in controlling fungal infections. Combining voriconazole with interferon gamma may be more effective than voriconazole alone in treating fungal infections.

PURPOSE: Randomized phase II trial to compare the effectiveness of voriconazole with or without interferon gamma in treating patients who have aspergillosis or other fungal infections.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety profile of voriconazole and interferon gamma in patients with invasive aspergillosis or other filamentous fungal infections.
* Compare the efficacy and possible heterogeneity in efficacy of voriconazole with or without interferon gamma across different patient sub-populations, in terms of designing a larger phase II or pivotal phase III study.
* Determine the time to partial or complete response and rate of response (at weeks 6 and 12 or at end of treatment and follow-up) in patients receiving interferon gamma.
* Compare the proportion of patients with at least a two-fold reduction in the galactomannan antigenemia titer at 6 and 12 weeks or at end of treatment with these regimens.
* Determine surrogate immunologic markers for response to interferon gamma, functional integrity and anti-fungal activity of phagocytic cells (neutrophils, monocytes, and macrophages), and nonphagocytic effector cells (natural killer and T cells) in these patients.

OUTLINE: This is a randomized, double-blind, multicenter, pilot study. Patients are stratified according to age (under 18 vs 18 and over) and absolute neutrophil count (less than 500/mm^3 vs at least 500/mm^3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive voriconazole (IV over 80-120 minutes for the first 3 doses and orally every 12 hours for subsequent doses) 3 times per week and interferon gamma subcutaneously (SC) 3 times per week.
* Arm II: Patients receive voriconazole as in arm I and placebo SC 3 times per week.

In both arms, treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 88 patients (44 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Proven or probable invasive aspergillosis or other filamentous fungal infection by cytology, histopathology, or culture within the past 7 days
* Presenting with 1 of the following:

  * Cancer
  * Aplastic anemia
  * Inherited immunodeficiencies
  * Autoimmune deficiency disorders
  * Acquired immunodeficiencies
  * Recipient of autologous peripheral blood stem cell or bone marrow transplantation
* CNS aspergillosis or other filamentous fungal infection allowed
* No invasive zygomycosis infection

PATIENT CHARACTERISTICS:

Age

* 2 and over

Performance status

* Not specified

Life expectancy

* At least 7 days

Hematopoietic

* Not specified

Hepatic

* ALT no greater than 5 times upper limit of normal

Renal

* Creatinine clearance at least 30 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No prior significant CNS disorder (e.g., multiple sclerosis or uncontrolled seizures)
* No prior grade 3 or 4 toxicity or severe allergic reaction to interferon gamma
* No prior intolerance or hypersensitivity to voriconazole or other azoles
* No acute or chronic graft-versus-host disease
* No conditions that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic peripheral blood or bone marrow transplantation
* No concurrent interferon alfa

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior solid organ transplantation

Other

* Prior voriconazole allowed
* At least 24 hours since prior administration of any of the following:

  * Astemizole
  * Cisapride
  * Pimozide
  * Quinidine
  * Sirolimus
  * Terfenadine
  * Rifabutin
  * Ergot alkaloids
  * Sildenafil citrate
  * Amiodarone
  * Flecainide
  * Systemic lidocaine
* More than 14 days since prior long-acting barbiturates, carbamazepine, or rifampin
* No other concurrent systemic antifungal drugs
* No other concurrent investigational agents

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-08; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Study Chair — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland